CLINICAL TRIAL: NCT03919266
Title: Combined Use of a Respiratory Broad Panel Multiplex PCR and Procalcitonin to Reduce Antibiotics Exposure in Adult Patients With Sickle-cell Disease Hospitalized for Acute Chest Syndrome. A Bi-centric, Open, Parallel-group, Randomized Controlled Study
Brief Title: Combined Use of a Respiratory Broad Panel Multiplex PCR and Procalcitonin to Reduce Antibiotics Exposure in Hospitalized Sickle-cell Adults With Acute Chest Syndrome.
Acronym: Antibio_STA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP180159
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Acute Chest Syndrome; Sickle Cell Disease
Keywords: Acute chest syndrome; SCD; PCR multiplex; antibiotic treatment
MeSH Terms: conditions — Acute Chest Syndrome; Anemia, Sickle Cell | interventions — Procalcitonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): usual antibiotic treatment
  Interventions: Procedure: Control: usual antibiotic treatment
- Intervention (Experimental): targeted antibiotic treatment according to the results of PCR multiplex
  Interventions: Procedure: Intervention: Combined use of a respiratory broad panel multiplex PCR and procalcitonin

INTERVENTIONS:
Procedure: Intervention: Combined use of a respiratory broad panel multiplex PCR and procalcitonin — The actions or procedures added by the research are the realization of a nasopharyngeal swab in the two strategies, and the PCT assay at D1, D3 and D7 in the pathogen-directed strategy
  Arms: Intervention
Procedure: Control: usual antibiotic treatment — usual antibiotic treatment
  Arms: Control

SUMMARY:
Many patients with Sickle Cell Disease (SCD) may develop Acute Chest Syndrome (ACS). ACS is usually caused by a Lower respiratory tract infection (LRTI) which may be caused by either a bacterium or a virus. Antibiotics are usually used for 7 to 10 days with no microbiological workup.

The hypothesis of the study is that the identification of the microorganisms might lead to a reduction of antibiotics exposure and a better care of the patients.

We speculate that an early pathogen-directed strategy (respiratory broad panel multiplex PCR and early antibiotics interruption based on the PCT values decrease) might reduce the antibiotics exposure in SCD patients with ACS who are hospitalized and for whom an antibiotic treatment is indicated, as compared with usual care

DETAILED DESCRIPTION:
Acute Chest Syndrome (ACS) is a frequent and severe acute complication of sickle-cell disease. It may affect 10 to 20% of hospitalized patients and is the leading cause of death. The symptoms combine a new pulmonary infiltrate and symptom(s) among fever, cough, dyspnea, expectoration, chest pain and crackles. The pathophysiology of ACS is complex and there are many interlinked aetiologies.

Lower respiratory tract infection (LRTI) is one of the most frequent aetiologies of ACS. Intracellular bacteria (Chlamydia, Mycoplasma), respiratory virus (especially respiratory syncytial virus) and pyogenes (Streptococcus pneumoniae and Staphylococcus aureus) are the most frequently identified microorganisms. Nevertheless, the clinical presentation of ACS is not helpful for the diagnosis of LRTI; the respiratory tract samples are not always collected, either because the patients do not expectorate or because the benefit-risk ratio of a fiberoptic bronchoscopy may be not advantageous. Moreover, usual diagnostic test are not enough performant.

The current practices rely on the systematic administration of antibiotics for 7 to 10 days. The efficacy and safety of alternative diagnostic and therapeutic strategies have never been evaluated in controlled clinical trial to cure ACS.

In this context, the optimisation of the microbiological documentation of ACS might enhance the use of antimicrobial drugs, reduce their duration, and limit the emergence of multidrug resistant bacteria.

Therefore, we speculate that an early pathogen-directed strategy (respiratory broad panel multiplex PCR and early antibiotics interruption based on the PCT values decrease) might reduce the antibiotics exposure in SCD patients with ACS who are hospitalized and for whom an antibiotic treatment is indicated, as compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Sickle Cell Disease patients with ACS with an antibiotic therapy indication
* Signed and informed consent
* Affiliated with social security

Exclusion Criteria:

Documented extra-pulmonary bacterial infection at the time of inclusion;

* Patients who received antibiotics for more than 24 hours before the diagnosis of ACS (during the primary hospitalization)
* Known severe immunosuppression (AIDS, neutropenia (<1000 PNN), hematology, solid tumor under chemotherapy, transplanted organ); long-term treatment with hydroxy-carbamide is not considered
* Pregnant or lactating women;
* Person deprived of liberty or under legal protection;
* Participation in another interventional study of type Jardé 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
to compare the antibiotics exposure at 28 days (D28) after the diagnosis of ACS between the two strategies | Day 28

SECONDARY OUTCOMES:
Rate of microbiological documentation of ACS | Day 28
Transfer to ICU at 28 days (D28) after the diagnosis of ACS between the two strategies | Day 28
Survival at 28 days | Day 28
occurrence of a secondary bacterial respiratory infection or any other secondary infection at 28 days | Day 28
Global use of antibiotics at 28 days | Day 28
Time to clinical stability at 28 days | Day 28
transfusion and exchange transfusion at 28 days | Day 28
ICU and hospital lengths of stay | Day 28
Readmission rate in hospital at 28 days | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Muriel FARTOUKH, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Réanimation et USC médico-chirurgicale, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sabate-Elabbadi A, Mekontso-Dessap A, Lionnet F, Santin A, Verdet C, Woerther PL, Lopinto J, Turpin M, Rousseau A, Lacoste-Badie R, Razazi K, Voiriot G, Fartoukh M. Combined use of respiratory multiplex PCR and procalcitonin to reduce antibiotic exposure in sickle-cell adult patients with acute chest syndrome (The ANTIBIO-STA study): a randomised, controlled, open-label trial. Lancet Reg Health Eur. 2025 Feb 7;51:101234. doi: 10.1016/j.lanepe.2025.101234. eCollection 2025 Apr. PMID 39995490